CLINICAL TRIAL: NCT07327671
Title: Developing and Efficiency Evaluation of a Positioning Assist Device for Urinary Catheterization in Female Patients
Brief Title: Positioning Device for Female Urinary Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Bircan Kolcak, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23232323
Record Dates: First submitted 2023-03-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2024-02

CONDITIONS: Urinary Catheterization; Device; Nursing; Positioning (Prone, Right Lateral and Semi-Elevated Supine Position); Randomised Controlled Trial
Keywords: urinary catheterization; assistive device; nursing; usebility testing; randomized cross-over trial; positioning device

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dorsal recumbent positioning device (Experimental): procedure performed with dorsal recumbent positioning device
  Interventions: Device: dorsal recumbent positioning device
- Control group (No Intervention)

INTERVENTIONS:
Device: dorsal recumbent positioning device — Participants in the supine positioning device group use this device prior to the procedure to ensure the supine position during urinary catheterisation in female patients. Once this device has safely secured the position, the steps for urinary catheterisation are carried out.
  Arms: dorsal recumbent positioning device

SUMMARY:
In female patients, the dorsal recumbent position is required to visualize the urethral meatus. In female patients, direct visualization of the urethral meatus after providing a suitable position is very important for successful catheter advancement while maintaining sterile conditions. Especially in unconscious or uncooperative female patients, it is much more difficult to maintain and maintain an appropriate position, and more than one staff may be needed for this. Although it is clear that it is important and difficult to position female patients during catheterization and maintain it throughout the procedure, no device used to assist positioning has been encountered. Therefore, in this project; The aim of this study is to provide a comfortable and safe position for the patient in urinary catheterization in female patients, to develop an auxiliary device to maintain this position throughout the procedure, and to evaluate the effectiveness of this device.

DETAILED DESCRIPTION:
Urinary elimination is one of the most fundamental physiological needs, and when it cannot be met by the individual for any reason, urinary catheterisation is required to drain urine accumulated in the bladder. Urinary catheterisation consists of a series of sequential steps. The first step is positioning the patient. In female patients, the dorsal recumbent position is required to visualise the urethral meatus. Once an appropriate position has been achieved in female patients, direct visualisation of the urethral meatus is crucial for the successful advancement of the catheter under sterile conditions. Providing and maintaining an appropriate position is particularly difficult in unconscious or uncooperative female patients, and may require multiple personnel. Although it is clear that positioning female patients during catheterisation and maintaining this position throughout the procedure is important and difficult, no devices have been found to assist with positioning. Therefore, this project aims to develop an assistive device to provide female patients with a comfortable and safe position during urinary catheterisation and to maintain this position throughout the procedure, and to evaluate the effectiveness of this device. To this end, a new positioning cushion will be developed, and a preclinical validation study will be conducted using a mixed-methods research design that includes a randomised controlled trial and a descriptive qualitative study.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse with at least a bachelor's degree
* Previous experience of urinary catheterization
* Having worked or working in intensive care
* Having voluntarily agreed to participate in the research

Exclusion Criteria:

* Leaving work voluntarily

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Urinary Catheterization Procedure Time (minutes) | From the start to the end of the catheterisation procedure, a maximum of 10 minutes
  Total time required to complete the urinary catheterization procedure, measured in minutes from video recordings, including preparation time, catheter insertion time, and total procedure duration.
Nurses' Lumbar Fatigue (Visual Analog Scale, VAS 0-100) | Day 1
  Lower back fatigue experienced by nurses during the procedure, assessed using a Visual Analogue Scale (VAS) from 0 to 100, where higher scores indicate greater fatigue.
Need for Support Personnel | Day 1
  Requirement for additional support staff during the procedure, recorded as yes/no based on video analysis.
Nurses' Physical Effort (Visual Analog Scale, VAS 0-100) | Day 1
  Physical effort perceived by nurses during the catheterization procedure, measured using a Visual Analogue Scale (VAS) from 0 to 100, where higher scores indicate greater physical effort.

SECONDARY OUTCOMES:
User Satisfaction (QUEST 2.0) | Day 1
  Satisfaction with the dorsal recumbent positioning device measured using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Gulhane Faculty of Nursing, Ankara, Turkey, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher-Gutowski S, Cecil J. Is 2-person urinary catheter insertion effective in reducing CAUTI? Am J Infect Control. 2019 Dec;47(12):1508-1509. doi: 10.1016/j.ajic.2019.05.014. Epub 2019 Jul 16. PMID 31324489
- [Background] Santos-Costa P, Alves M, Sousa C, Sousa LB, Paiva-Santos F, Bernardes RA, Ventura F, Salgueiro-Oliveira A, Parreira P, Vieira M, Graveto J. Nurses' Involvement in the Development and Usability Assessment of an Innovative Peripheral Intravenous Catheterisation Pack: A Mix-Method Study. Int J Environ Res Public Health. 2022 Sep 5;19(17):11130. doi: 10.3390/ijerph191711130. PMID 36078842
- See also: Urinary Catheter Care Guidelines Version: 6 — https://www.scribd.com/document/818158489/Urinary-Catheter-Guidelines-V6